CLINICAL TRIAL: NCT03221179
Title: A Randomized, Adaptive, Investigator/ Subject Blind, Single Ascending Dose, Placebo-Controlled Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered RO7049665 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7049665 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: WP39826
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RO7049665 (Experimental): Participants will be administered a single SC dose of RO7049665 administered in up to 4 SC injection.
  Interventions: Biological: RO7049665
- Placebo (Placebo Comparator): Participants will be administered a single SC dose of matching placebo formulation administered in up to 4 SC injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RO7049665 — A single ascending dose (starting dose 1.5 micrograms [mcg])of RO7049665 will be administered SC.
  Arms: RO7049665
Biological: Placebo — Matching placebo will be administered SC once.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single ascending doses of subcutaneous (SC) injections of RO7049665 in healthy volunteers. In addition, pharmacokinetics (PK) of RO7049665, the effects of single doses of RO7049665 on regulatory T-cells as well as the single dose immunogenicity of RO7049665 will be evaluated. This trial plans to evaluate approximately seven single dose-levels of RO7049665 or matching-placebo during dose-escalation in approximately 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers, 18 to 45 years of age, inclusive;
* Absence of evidence of any active or chronic disease;
* Body mass index (BMI) of 18-30 kilograms per square meter (kg/m^2), inclusive;
* Contraception requirements: refrain from heterosexual intercourse or use contraceptive measures, and agreement to refrain from donating sperm.

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis;
* Clinically significant abnormalities (as judged by the Investigator) in laboratory test results;
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study;
* History of hypersensitivity to biologic agents or any of the excipients in the formulation;
* Any abnormal skin conditions or potentially obscuring tattoos, pigmentation or lesions in the area intended for subcutaneous injection;
* Prior administration of aldesleukin, or interleukin-2 (IL-2) derivatives.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From baseline up to approximately 8 weeks
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

SECONDARY OUTCOMES:
PK: Time to Maximum Concentration (Tmax) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum and the time from SC injection to maximum concentration of RO7049665 will be determined.
PK: Maximum Serum Concentration Observed (Cmax) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum and the maximum concentration of RO7049665 will be determined.
PK: Area Under the Concentration-Time Curve (AUC) from Time 0 to Time of Last Sampling of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. AUC from time of drug administration to last blood sampling (AUClast) will be determined in a plot of RO7049665 serum concentration versus time.
PK: AUC from Time 0 to infinity (AUCinf) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. AUC from time of drug administration extrapolated to infinity (AUCinf) will be determined in a plot of RO7049665 serum concentration versus time.
PK: AUC from Time 0 to Time tau (AUC0-t) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. AUC from time of drug administration to time tau (AUC0-t), which is defined as the time of last measurable serum concentration, will be determined in a plot of RO7049665 serum concentration versus time.
PK: Apparent Clearance (CL/F) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. Clearance, which is a measure of the rate at which a drug is metabolized or eliminated, will be determined.
PK: Apparent Volume of Distribution (Vz/F) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. Volume of distribution of RO7049665 will be determined.
PK: Half-life (t1/2) of RO7049665 | Pre-dose on Day 1, post-dose on Day 1 at 2 hours (h), 6 h and 12 h, once daily on Days 2-8, Day 12, Day 15, Day 21, Day 29 and Day 43
  Blood samples will be taken pre-dose and at multiple time points after dose administration. RO7049665 concentration will be analyzed in serum. t1/2 is the time required for the serum concentration of RO7049665 to be reduced to half.
Change from Baseline in Regulatory T Lymphocyte (Tregs) Count | Day -1, Pre-dose Day 1; post-dose Day 2, 3, 4, 6, 8, 12, 15, 29, up to follow-up visit (Day 57)
  Blood samples will be taken for flow cytometry and peripheral blood mononuclear cell (PBMC) isolation. Markers for quantification of Tregs will be assessed.
Percentage of Participants with Anti-Drug Antibodies | Pre-dose Day 1, post-dose Day 8, 15, 29, up to follow-up visit (Day 57)
  Anti-drug antibody assays will be used to detect anti-drug antibodies against RO7049665. Samples which are positive for anti-drug antibodies will be further assessed using a neutralizing antibody assay.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences Early Development Services, Zuidlaren, Netherlands